CLINICAL TRIAL: NCT02464748
Title: Telehealth in Motor Neurone Disease: A Single Centre, Randomised Controlled Feasibility and Pilot Study of the Use of the TiM Telehealth System to Deliver Highly Specialised Care in Motor Neurone Disease at a Distance
Brief Title: Telehealth in Motor Neurone Disease
Acronym: TiM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17165; 26675465 (Registry Identifier: ISRCTN); 17022 (Registry Identifier: National Institute for Health Research Portfolio ID)
Record Dates: First submitted 2014-11-13; First posted 2015-06-08 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Motor Neuron Disease
MeSH Terms: conditions — Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients and their primary carer will use a weekly telehealth system. This involves a series of questions on a tablet computer that is transmitted to their regional MND care centre for review and action.
  Interventions: Other: TiM telehealth arm
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: TiM telehealth arm
  Arms: Intervention

SUMMARY:
Motor neurone disease (MND) is a rare but debilitating neurological condition that causes paralysis of the body's muscles leading to severe disability and eventually death. Patients often struggle to travel the long distances to specialist clinics to receive the care they require whilst this expert care is often unavailable in the community. Telehealth has the potential to enable a specialist team to monitor the health and wellbeing of patients and their carers whilst they are at home. This could improve the patient's health, improve the quality of life of both patients and their carers, and lead to more effective use of health resources.

This is a randomised controlled pilot study that will involve 40 patients who are cared for by the Sheffield Motor Neurone Disease care centre and their main informal carer (a total of 80 participants). Half of the participants will use the telehealth system for a minimum of six months and maximum of eighteen months and information will be collected from patients, carers and their care team. This will include collecting clinical outcome measures, health resource use and the opinions and experience of using the system. All participants will continue to receive their usual care.

This is a pilot study. It aims to determine the feasibility and acceptability of the telehealth system to patients, carers and their health care providers. It also aims to determine how a larger trial could successfully evaluate the clinical and cost-effectiveness of the system.

DETAILED DESCRIPTION:
MND is often referred to as amyotrophic lateral sclerosis (ALS) or Lou Gehrig's disease.

ELIGIBILITY:
Patient Inclusion Criteria:

* Patients aged 18 years or over who have attended the MND clinic at the Royal Hallamshire Hospital, Sheffield.
* Patients with amyotrophic lateral sclerosis diagnosed by a consultant neurologist with symptom onset within the last three years.

  o Or
* Patients with amyotrophic lateral sclerosis, primary muscular atrophy or progressive lateral sclerosis diagnosed by a consultant neurologist with a deterioration in their condition as evidenced by a deterioration in the ALS functional rating score (ALSFRS-R) by at least two points during the previous 18 months.
* Live within 120 minute drive from Sheffield

Patient Exclusion Criteria:

* Patients attend another MND care centre in the UK.
* Significant impairment in decision making capacity preventing informed consent by the subject due to a major mental disorder including fronto-temporal dementia.
* Patient unable to use the TiM system due to physical, intellectual or language difficulties and unwilling to permit carer to operate it on their behalf. Patients will be asked to complete two questions used within the TiM system, with, or without the help to their carer to verify their ability to use the system.
* The patient has no eligible informal carer willing to participate in the trial
* Insufficient mobile telephone reception in the patients' home to use the TiM system.
* Any other major impairment that may affect their ability to participate in the study

Carer inclusion criteria

* Age 18 years or older
* Person identified by the patient as the major provider of informal care (emotional and/or practical support) to the patient and provides more than one hour per week of unpaid care
* Carer willing to allow data they provide during the trial to be shared by the research team with their own doctor in the event of serious clinical need.

Carer exclusion criteria

* Significant decision making capacity preventing informed consent due to a major mental disorder.
* Carer unable to use the TiM system due to physical, intellectual or language difficulties. Carers will be asked to complete two questions used within the TiM system to verify their ability to use the system.
* Inability to participate in the study due to other major physical or mental illness or language difficulties.
* Professional carers receiving direct payment for their services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of using the telehealth system from interviews | Up to 18 months
  Recruitment rate, retention rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Institute for Translational Neurosciences, Sheffield, United Kingdom